CLINICAL TRIAL: NCT01824225
Title: Study of PRN and Every 2months Intravitreal Aflibercept After 3 Initial Monthly Injection for Age Related Macular Degeneration
Brief Title: Study of PRN and Every 2months Intravitreal Aflibercept for Age Related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Koji Tanaka, Lecturer, Nihon University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NihonU-2
Record Dates: First submitted 2013-03-31; First posted 2013-04-04 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Age-related Macular Degeneration
Keywords: aflibercept; intravitreal injection
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRN injection of aflibercept (Active Comparator): Intravitreal aflibercept
  Interventions: Drug: Aflibercept
- Two months injection of aflibercept (Active Comparator): Intravitreal afilibercept
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept

SUMMARY:
Evaluate a treatment result of every two months versus as needed (PRN) after 3 initial monthly intravitreal aflibercept for the Japanese age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of age-related macular degeneration

Exclusion Criteria:

* Any treatment before intravitreal Aflibercept for age-related macular degeneration.
* Visual acuity above 0.1 in decimal visual acuity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Visual acuity after treatment by PRN or 2 months intravitreal Aflibercept | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuko Yuzawa, M.D., Study Chair — Surugadai Nihon University Hospital
Locations (1):
- Surugadai Nihon university hospital, Chiyoda-ku, Tokyo, Japan